CLINICAL TRIAL: NCT05188092
Title: Effect of Lung Ultrasound-Guided Fluid Deresuscitation on Duration of Ventilation in Intensive Care Unit Patients (CONFIDENCE)
Brief Title: Lung Ultrasound-Guided Fluid Deresuscitation in ICU Patients
Acronym: CONFIDENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. Dr. M.J. Schultz, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONFIDENCE
Record Dates: First submitted 2021-12-22; First posted 2022-01-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Mechanical Ventilation; Fluid Overload; Deresuscitation; Ventilator-free Days
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Routine fluid deresuscitation in which fluid withdrawal is started and continued at the discretion of the treating physician.
- Intervention (Active Comparator): Deresuscitation is guided by lung ultrasound observations.
  Interventions: Other: Lung ultrasound guided deresuscitation

INTERVENTIONS:
Other: Lung ultrasound guided deresuscitation — With every new LUS examination, the following scenarios, with distinct recommendations, are possible:
  1. LUS observations suggest massive pulmonary fluid overload, with the recommendation to minimize fluid infusion and start fluid withdrawal, targeting a negative fluid balance of at least -1500 ml in the next 24 hours;
  2. LUS suggests some pulmonary edema and/or significant pleural effusion. These LUS observations suggest little pulmonary fluid overload, with the suggestion to minimize fluid infusion and start fluid withdrawal, targeting a negative fluid balance at least -500 ml in the next 24 hours;
  3. LUS suggests absence of pulmonary edema and no pleural effusion. These LUS observations suggest no fluid overload, with the suggestion to target a neutral fluid balance in the next 24 hours.
  Arms: Intervention

SUMMARY:
Timely recognition and treatment of fluid overload can expedite liberation from invasive mechanical ventilation in intensive care unit (ICU) patients. Lung ultrasound (LUS) is an easy to learn, safe, cheap and noninvasive bedside imaging tool with high accuracy for pulmonary edema and pleural effusions in ICU patients. The aim of this study is to assess the effect of LUS-guided deresuscitation on duration of invasive ventilation in ICU patients. The investigators hypothesize that LUS-guided fluid deresuscitation is superior to routine fluid deresuscitation (not using LUS) with regard to duration of invasive ventilation.

This study is an international multicenter randomized clinical trial (RCT) in invasively ventilated ICU patients.This study will include 1,000 consecutively admitted invasively ventilated adult ICU patients, who are expected not to be extubated within the next 24 hours after randomization. Patients are randomly assigned to the intervention group, in which fluid deresuscitation is guided by repeated LUS, or the control group, in which fluid deresuscitation is at the discretion of the treating physician (not using LUS).

DETAILED DESCRIPTION:
Objective:

The aim of this study is to assess the effect of LUS-guided deresuscitation on duration of invasive ventilation in ICU patients.

Hypothesis:

LUS-guided fluid deresuscitation is superior to routine fluid deresuscitation (not using LUS) with regard to duration of invasive ventilation.

Study design:

The CONFIDENCE study is an investigator-initiated, national, multicenter, randomized clinical trial in critically ill invasively ventilated patients admitted to the ICUs of participating hospitals.

Study population:

Adult patients admitted to ICUs in multiple countries

Sample size calculation:

The sample size is computed on the basis of the hypothesis that LUS guided deresuscitation is associated with a reduction of two days of ventilation. Assuming a mean (±SD) number of VFD-28 of 13±11 days, the ivenstigators estimate that a sample of 1000 patients (500 per group) is needed to have 80% power, at a two-tailed significance level of 0.05, to detect a mean between-group difference of 2 VFD-28, and allowing an anticipated dropout rate of 5%.

Methods:

Patients in participating intensive care units (ICU) are screened for eligibility. Inclusion and randomization will occur within 24 hours after meeting the inclusion criteria. If possible, informed consent from the legal representative will be obtained before randomization but no longer than 48 hours after meeting the inclusion criteria.

Patients are eligible if they are admitted to one of the participating ICUs, are invasively ventilated for less than 24 hours at randomization and expected to be under invasive ventilation for longer than 24 hours after randomization.

Randomization will be performed using Castor Electronic Data Capture (EDC). A dedicated, password protected, encrypted website. Randomization sequence is generated by a dedicated computer randomization software program. Due to the nature of the intervention, blinding of the caregivers is not possible.

Patients will be randomly assigned in a 1:1 ratio to lung guided fluid deresuscitation or routine fluid deresuscitation. Randomization will be stratified per center.

Lung ultrasound guided deresuscitation: with lung ultrasound (LUS)-guided fluid deresuscitation, LUS examinations are performed at least onze a day in hemodynamically stable patients, defined as a mean arterial pressure (MAP) ≥ 65 mmHg (with vasopressor dose decreasing and norepinephrine ≤ 0.2 μg/kg/min), and no new clear signs of hypoperfusion such as mottled skin and capillary refill time > 3 seconds and/or new oliguria (urine output < 0.3-0.5ml/kg/hour for the previous 6 hours). Target MAP can be changed in conditions in which 65 mmHg is not sufficient (i.e. history of chronic hypertension). In these cases the target MAP is at the discretion of the treating physician. 12-region LUS is performed, by a trained healthcare provider, and each region is scanned for the presence of B-lines and pleural effusions and scored using the lung ultrasound score. After extubation, lung ultrasound is continued once a day until day 28 or until discharge (whatever comes first) to monitor reappearance of pulmonary fluid overload or pleural effusion. In case of reappearance (or increase) of pulmonary fluid overload or pleural effusion, fluid withdrawal is started again according to the treatment protocol.

Routine deresuscitation: in routine fluid deresuscitation, in which fluid withdrawal is started and continued at the discretion of the treating physician, factors guiding fluid deresuscitation are chosen by the treating physician and may include the following: physical examination, laboratory values (e.g. BNP), chest x-ray, PiCCO or pulmonary artery catheters. LUS examinations are not performed to guide fluid deresuscitation in this group.

In both groups patients are extubated if standard extubation criteria are fulfilled, i.e., normal body temperature, patient awake and responsive/cooperative, adequate cough reflex, adequate oxygenation and ventilation, and hemodynamically stable.

Monitoring:

Monitoring of patients safety and reviewing of safety issues is performed by a designated independent Data Safety and Monitoring Board (DSMB).The DSMB watches over the ethics of conducting the study in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Admission to one of the participating ICUs;
* Invasively ventilated for less than 24 hours at randomization;
* Expected to be under invasive ventilation for longer than 24 hours after randomization.

Exclusion Criteria:

* Age below 18 years old;
* Suspected or confirmed pregnancy;
* Participation in other interventional trials with similar endpoints;
* Use of long term home mechanical ventilation;
* Neurological condition that can prolong duration of mechanical ventilation (i.e.Guillain-Barré syndrome, high spinal cord lesion, amyotrophic lateral sclerosis, multiple sclerosis, or myasthenia gravis);
* Conditions in which LUS cannot be performed or correctly interpreted (i.e. chest wall abnormalities, morbid obesity, and pre-existing interstitial lung disease);
* Conditions in which targeting a negative fluid balance is discouraged (i.e. subarachnoid bleeding, severe rhabdomyolysis (CK > 20.000);
* Previous participation in this RCT;
* Patients transferred from another center and invasively ventilated for longer than 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Ventilator free days(VFD) and alive at day 28 | 28 days after randomisation
  Patient is alive and breathes without assistance of the mechanical ventilator, if the period of unassisted breathing lasted at least 24 consecutive hours:
  * VFD-28 = 0 if subject dies within 28 days of mechanical ventilation
  * VFD-28 = 28 - x if successfully liberated from ventilation x days after initiation Succcessful liberation: extubation (planned or unplanned) without death or reintubation within the next 72 hours
  * VFD-28 = 0 if the subject is mechanically ventilated for ≥ 28 days

SECONDARY OUTCOMES:
Duration of ventilation | 28 days
  Duration of ventilation in survivors
ICU length of stay | 28 days
  Length of stay in the intensive care unit
Hospital length of stay | 28 days
  Length of stay in the hospital
28 day mortality | 28 days
  Mortality after 28 days
90 day mortality | 90 days
  Mortality after 90 days
Incidences of reintubations | 28 days
  Need of reintubation within 72 hours after extubation
Cumulative fluid balances after randomization | 7 days
  Cumulative fluid balance on day 1-7 after randomization;
Cumulative fluid balances after start of lung ultrasound examination | 7 days
  Cumulative fluid balance on day 1-7 after start of lung ultrasound examinations;
Incidence of acute kidney injury | 28 days
  Kidney injury with Kidney Disease Improving Global Outcomes (KDIGO) stadium ≥ 2

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J Schultz, Prof, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Pieter Roel Tuinman, Dr, Principal Investigator — Amsterdam UMC, location VUmc; Frederique Paulus, Dr, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Leo MA Heunks, Study Director — Amsterdam UMC, location VUmc
Locations (3):
- Netherlands (3):
  - Rijnstate, Arnhem, Gelderland
  - Amsterdam UMC, location VUMC, Amsterdam, North Holland
  - Amsterdam UMC, location AMC, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Blok SG, Mousa A, Brouwer MG, de Grooth HJ, Neto AS, Blans MJ, den Boer S, Dormans T, Endeman H, Roeleveld T, Scholten H, van Slobbe-Bijlsma ER, Scholten E, Touw H, van der Ven FSLIM, Wils EJ, van Westerloo DJ, Heunks LMA, Schultz MJ, Paulus F, Tuinman PR. Effect of lung ultrasound-guided fluid deresuscitation on duration of ventilation in intensive care unit patients (CONFIDENCE): protocol for a multicentre randomised controlled trial. Trials. 2023 Mar 24;24(1):226. doi: 10.1186/s13063-023-07171-w. PMID 36964614

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-11-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT05188092/SAP_000.pdf